CLINICAL TRIAL: NCT01177267
Title: Prevalence of Potential Cytochrome P450 Pharmacokinetic Incident Drug-Drug Interactions Among Osteoarthritis Patients Taking Opioid Analgesics and Associated Economic Outcomes
Brief Title: Prevalence of Potential Cytochrome P450 Pharmacokinetic Incident Drug-Drug Interactions(DDI) Among Osteoarthritis Patients
Status: Completed | Type: Observational
Sponsor: NEMA Research, Inc. (Industry)
Responsible Party: Principal Investigator, Joseph Pergolizzi, MD, Principal Investigator, NEMA Research, Inc.
Other Study IDs: CYP450OA3
Record Dates: First submitted 2010-08-05; First posted 2010-08-06 (Estimated); Last update posted 2012-05-01 (Estimated); Status verified 2012-04

CONDITIONS: Osteoarthritis
Keywords: retrospective database analysis in osteoarthritis patients
MeSH Terms: conditions — Osteoarthritis

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: Yes

SUMMARY:
Using a retrospective database analysis, OA patients taking at least one CYP450-metabolized opioid (codeine, fentanyl, hydrocodone, methadone, oxycodone, or tramadol) and at least one other prescription drug metabolized via the CYP450 system were evaluated for an incident drug-drug exposure (DDE), which places them at risk for experiencing a pharmacokinetic drug-drug interaction (DDI).

ELIGIBILITY:
Inclusion Criteria:

* osteoarthritis

Exclusion Criteria:

* pregnancy

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: retrospective database analysis
Sampling Method: Non-Probability Sample
Enrollment: 10000
Dates: Start 2010-09; Primary Completion 2010-12 (Actual); Study Completion 2011-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Joseph Pergolizzi, MD, Principal Investigator — NEMA Research